CLINICAL TRIAL: NCT02932345
Title: A Study of Clinical and Genomic Analysis on Long-term Survivors of EGFR Mutation Positive Advanced Non-small-cell Lung Cancer Patients With Gefitinib Treatment in China
Brief Title: Gefitinib Long-term Survivor Study
Status: Terminated | Type: Observational
Why Stopped: Due to strategic decision, AZ has applied to terminate study at all participating sites and has committed that the data generated during the course of the study will not be submitted to China National Medical Products Administration.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7913R00020
Record Dates: First submitted 2016-09-12; First posted 2016-10-13 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2021-12

CONDITIONS: EGFR Mutation Positive Advanced Non-small-cell Lung Cancer
Keywords: EGFR mutation; non-small-cell lung cancer;
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Long-term survivors group (case): EGFR M+ aNSCLC patients who continuously received gefitinib for at least 3 years
- Rapid PD group (control): EGFR M+ aNSCLC patients who had undergone PD after gefitinib treatment≤3 months

SUMMARY:
The primary objective is to describe the genomic profile of long-term survivors, especially to find out potential genomic prognosis and/or predictive factors for gefitinib long-term efficacy as compared to rapid PD patients

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the long-term survivors group, the study subjects must fulfil the following criteria at the time of screening:

1. Provision of informed consent or EC approve informed consent waiver prior to any study specific procedures
2. Histological or cytological confirmed locally advanced NSCLC (stage III B) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy
3. EGFR mutation positive
4. Patients who continuously received gefitinib for at least 3 years without evidence of PD
5. Patients with OS ≥ 5 years from NSCLC diagnosis will be preferred
6. Collect archival tumour tissue before gefitinib treatment (blood and re-biopsy tumour tissue are optional); tumor tissue samples requirements: 1) slices requirements: >1 cm2, thickness 4-5 μm, ≥ 15 slices. or, whole FFPE block; 2) tumor percentage > 20% and necrosis < 30% by pathology QC.

For inclusion in the rapid PD group, the study subjects must fulfil the following criteria:

1. Provision of informed consent or EC approve informed consent waiver prior to any study specific procedures
2. Histological or cytological confirmed locally advanced NSCLC (stage III B) or metastatic (stage IV) NSCLC, not amenable to curative surgery or radiotherapy
3. EGFR mutation positive
4. Patients who had undergone PD after gefitinib treatment≤3 months (Rapid PD)
5. Collect archival tumour tissue before gefitinib treatment (blood and re-biopsy tumour tissue samples are optional) ; tumor tissue samples requirements: 1) slices requirements: >1 cm2, thickness 4-5 μm, ≥ 15 slices. or, whole FFPE block; 2) tumor percentage > 20% and necrosis < 30% by pathology QC.

Exclusion Criteria:

For the active patients, who must not enter the study if any of the following exclusion criteria are fulfilled 1. Patients who disagree to participate this study.

For the terminated patients, who must not enter the study if any of the following exclusion criteria are fulfilled

1. Patients in whose medical objection was recorded to use the existing data from medical practice for scientific research.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will recruit approximately 150 aNSCLC patients who fulfil the inclusion/exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2016-10-31 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with specific genomic alterations(mutation, copy number change and fusion) of short or long-term survivors | at time of sample collection before Gefitinib treatment initiation, up to 10 years before study start

SECONDARY OUTCOMES:
Sex | at time of Gefitinib treatment initiation,up to 10 years before study start
Age | at time of Gefitinib treatment initiation, up to 10 years before study start
Pre-existing comorbidities at initiation of gefitinib therapy | at time of Gefitinib treatment initiation, up to 10 years before study start
Cancer type and date of first ever cancer diagnosis | at time of Gefitinib treatment initiation, up to 10 years before study start
Histological subtype | at time of Gefitinib treatment initiation, up to 10 years before study start
Location(s) of metastatic disease at initiation of gefitinib therapy for subjects with TNM stage IV disease | at time of Gefitinib treatment initiation, up to 10 years before study start
EGFR mutation status | at time of Gefitinib treatment initiation, up to 10 years before study start
Smoking status | at time of Gefitinib treatment initiation, up to 10 years before study start
ECOG performance status at time of Gefitinib treatment initiation | at time of Gefitinib treatment initiation, up to 10 years before study start
Gefitinib treatment patterns- Starting dose | at time of Gefitinib treatment initiation, up to 10 years before study start
Gefitinib treatment patterns- Dose reductions, treatment interruptions, discontinuation including reasons | from Gefitinib treatment initiation to Gefitinib treatment discontinuation or study completion, whichever occurred first, up to 12 years
Gefitinib treatment patterns- Types of other systemic therapies given in combination with gefitinib | from Gefitinib treatment initiation to Gefitinib treatment discontinuation or study completion, whichever occurred first, up to 12 years
Therapeutic agent name post-gefitinib discontinuation | from gefitinib discontinuation to one year post- gefitinib discontinuation, around one year
Documented tumour response (complete or partial response or stable disease, according to RECIST) as determined by the treating physician by clinical judgment and/or imaging after first ever initiation of gefitinib | from Gefitinib treatment initiation to study completion, up to 12 years
Progression Free Survival (PFS) | from Gefitinib treatment initiation to disease progression or study completion, whichever occurred first, up to 12 years
Overval survival (OS) | from Gefitinib treatment initiation to death or study completion, whichever occurred first, up to 12 years

CONTACTS AND LOCATIONS:
Overall Officials: Yilong WU, Professor, Principal Investigator — Guangdong Provincial People's Hospital
Locations (14):
- China (14):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Xi'an, Shaanxi
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Taiyuan, Shanxi
  - Research Site, Chengdu, Sichuan
  - Research Site, Hangzhou, Zhejiang